CLINICAL TRIAL: NCT03042689
Title: Phase I Study of Regorafenib in Patients With Advanced Myeloid Malignancies
Brief Title: Study of Regorafenib in Patients With Advanced Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Gabriela Hobbs, Gabriela Hobbs, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-464
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib will be administered on a 28 day cycle Treatment will be administered on outpatient basis at a pre-determine dosage.
  Other Names: Stivarga

SUMMARY:
This research study is studying a drug as a possible treatment for advanced myeloid malignancies including AML (acute myeloid leukemia), MDS (myelodysplastic syndrome) and MPN (myeloproliferative neoplasms)

The intervention involved in this study is:

-Regorafenib (Stivarga)

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Regorafenib for this specific disease but it has been approved for other uses.

In this research study, the investigators are looking for the best dose of Regorafenib to treat the participant's disease with. Researchers will also look at how effective the study drug is in treating the participant's disease and if any side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed/refractory advanced malignancies. Specifically: relapsed refractory refractory acute myeloid leukemia that have failed one line of prior therapy, myelodysplastic syndrome that have failed hypomethylating agents, myelofibrosis that have failed ruxolitinib or are ineligible for this therapy.
* 18 years of age or greater.
* ECOG performance status of 0-1.
* Able to provide informed consent.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Able to swallow and retain oral medication.
* Normal organ and marrow function defined as:

  * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN) except for patients with Gilbert's disease.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer).
  * Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver or bone involvement of their cancer).
  * Serum creatinine ≤ 1.5 x the ULN.
  * International normalized ratio (INR)/ Partial thromboplastin time (PTT) ≤ 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists.)

Exclusion Criteria:

* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter the study.
* Systemic antineoplastic therapy in the past 14 days (excluding hydroxyurea).
* Uncontrolled hypertension (systolic pressure >140 mmHg or diastolic pressure > 90 mmHg on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > Class II.
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Eligible for, have a suitable donor and are willing to undergo Hematopoietic Stem Cell Transplantation (HSCT)
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Thrombotic, embolic, venous or arterial events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months of informed consent.
* Previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated non-melanoma skin carcinoma, noninvasive aerodigestive neoplasms or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed. All cancer treatments must be completed at least 3 years prior to registration.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Presence of a non-healing wound, non-healing ulcer or bone fracture.
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication.
* Renal failure requiring hemo-or peritoneal dialysis.
* Seizure disorder requiring medication.
* Persistent proteinuria ≥ Grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant). Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding, or intend to become pregnant during the study. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Presence of unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 grade 0 or 1 with the exception of alopecia. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by regorafenib (e.g. hearing loss, neuropathy) may be included after consultation with the principal investigator.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of regorafenib in patients with advanced myeloid malignancies | 2 years
  To determine the maximum tolerated dose regorafenib in patients with advanced myeloid malignancies.

SECONDARY OUTCOMES:
Pharmacodynamic effects of regorafenib on cell signaling pathways | 2 years
  To assess pharmacodynamic effect of regorafenib on cell signaling pathways such as FLT-3, RAS and other specific mutations found in each patient's leukemia.
Progression Free Survival | 2 years
Overall Survival | 2 years
To Measure Changes In Specific Markers Of Allele Burden | 2 years
  Measure changes in allele burden with regorafenib treatment using next generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No